CLINICAL TRIAL: NCT04708275
Title: A Waitlist Controlled Trial for Early Childhood Depression
Brief Title: Treatment of Early Childhood Depression
Acronym: PaCT_RCTwait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Lars White, Coordinating Investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-WAIT-SAD-KIDS
Record Dates: First submitted 2020-02-24; First posted 2021-01-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: Early Childhood Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: 2 arms, waitlist-controlled, randomized, single masked (outcomes assessor), single-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PaCT (Experimental): Manualized Psychoanalytic short-term therapy (PaCT) for children with internalizing disorders, 20-25 sessions (1, 2). PaCT helps the child to resolve rigid conflictual internal representations/ working models by using interpretative and mentalizing techniques and drawing on therapeutic transference relationship with the child and the parent.
  Interventions: Procedure: PaCT
- Waitlist (Active Comparator): PaCT after a waiting period (3 months)
  Interventions: Procedure: PaCT

INTERVENTIONS:
Procedure: PaCT — Manualized Psychoanalytic short-term therapy (PaCT) for children with internalizing disorders, 20-25 sessions (1, 2). PaCT helps the child to resolve rigid conflictual internal representations/ working models by using interpretative and mentalizing techniques and drawing on therapeutic transference relationship with the child and the parent.

SUMMARY:
Depression often occurs in early childhood. Moreover, later depression is frequently preceded by early childhood Depression (ECD). However, at present, there is a lack of evidence-based tratestments (EBTs) for ECD, posing a core research desideratum highlighted by both the American and German practice parameters for ECD. The current study seeks to redress this research gap, by evaluating the feasibility and dose-dependent effectiveness of manualized short-term psychoanalytic child psychotherapy (PaCT) compared to waitlist in a randomized controlled trial (RCT) among clinically referred 3 to 8-year-olds with ECD. Comprising 20-25 sessions in alternating settings (child-only, caregiver(s)-child, caregiver(s)-only), PaCT focuses on internal conflicts and representations underlying depressive disorders. PaCT targets the child-therapist relationship, using interpretative, play and mentalization-based techniques, aiming to elicit the interpersonal meaning of the child's symptoms within the child-caregiver relationship(s).

DETAILED DESCRIPTION:
For this trial, 62 clinically referred children meeting criteria for DSM-5 depressive disorders, will be randomized randomized to PaCT (n=31) or waitlist (n=31). The overarching aim is to engender reduction in depressive symptoms and diagnoses following PaCT vs. waitlist in order to determine effect sizes which can be used in power calculations for future large-scale clinical trials. Moreover, effects of PaCT will also be examined at mid-treatment to provide a first insight into the necesary therapeutic dose. Moreover, the trial will also be used as a first opportunity to examine feasibility of PaCT in young children, treatment integrity, as well as treatment acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 8 years
* DSM-5 depressive disorder (Major Depression, Dysthymia, Depression NOS), adapted for young children according to the AACAP criteria
* Written informed consent of patient's parents or guardian
* informed verbal assent from children (age >= 6 years)

Exclusion Criteria:

* IQ < 70
* autism spectrum or schizophrenia spectrum disorder in the child
* insufficient German language skills to participate in treatment (child or caregiver)
* ongoing litigation regarding child custody
* concurrent intensive psychotherapy
* participation in other interventional trials
* suspected lack of compliance

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Sum of depressive symptoms as indexed by the Preschool Age Psychiatric Assessment (PAPA) interview with the primary caregiver | post-treatment (after 20-25 weeks with weekly treatment sessions; on average after 7 months)
  Sum of depressive symptoms using Preschool Age Psychiatric Assessment (PAPA) at post-treatment in the treatment group compared to post-waiting period in the waitlist group (controlling for the respective pre-values) based on clinical interviews. The scale ranges from 0-9 symptoms and higher values indicate worse outcome.

SECONDARY OUTCOMES:
Sum of PAPA depressive symptoms | mid-treatment (after 12 weeks with weekly treatment sessions) and follow up (3 months after intervention)
  Sum of depressive symptoms using the PAPA. The scale ranges from 0-9 symptoms and higher values indicate worse outcome.
Diagnosis of depression | mid-treatment (after 12 weeks with weekly treatment sessions) and follow up (3 months after intervention)
  occurrence of diagnosis of depression using PAPA
Diagnosis of anxiety disorder | pre-waitlist (before waiting period) / pre-treatment (within 3 weeks before start of intervention), post-treatment (after 20-25 weeks with weekly treatment sessions) and follow up (3 months after intervention)
  occurrence of diagnosis of anxiety disorder using PAPA
Teacher-reported internalizing symptoms (TRF) | pre-waitlist (before waiting period)/pre-treatment (within 3 weeks before start intervention)/mid-treatment (after 12 weeks with weekly treatment sessions)/post-treatment (after 20-25 weeks with weekly treatment sessions)/FUP (3 months post intervention)
  (Nursery-)teacher-rated internalizing symptoms using Teacher Report Form (TRF). The scale ranges from 0-70 with higher scores indicating worse outcomes.
Interview-based internalizing symptoms | pre-waitlist (before waiting period), pre-treatment (within 3 weeks before start intervention), post-treatment (after 20-25 weeks with weekly treatment sessions), follow-up (3 months after intervention)
  Child self-reported internalizing symptoms using Berkeley Puppet Interview, the scale ranges from 1-182 with higher scores indicating better outcomes.
Caregiver-reported externalizing symptoms | pre-waitlist (before waiting period)/pre-treatment (within 3 weeks before start intervention)/mid-treatment (after 12 weeks with weekly treatment sessions)/post-treatment (after 20-25 weeks with weekly treatment sessions)/FUP (3 months post intervention)
  Externalizing symptoms rated by caregiversusing Child Behavior Checklist. (CBCL 4-18) The scale ranges from 0-66 with higher scores indicating worse outcomes.
Teacher-reproted externalizing symptoms | pre-waitlist (before waiting period)/pre-treatment (within 3 weeks before start intervention)/mid-treatment (after 12 weeks with weekly treatment sessions)/post-treatment (after 20-25 weeks with weekly treatment sessions)/FUP (3 months post intervention)
  Externalizing symptoms rated by teachers using Teacher Report Form (TRF). The scale ranges from 0-68 with higher scores indicating worse outcomes.
Cortisol secretion | pre-waitlist (before waiting period)/pre-treatment (within 3 weeks before start intervention)/mid-treatment (after 12 weeks with weekly treatment sessions)/post-treatment (after 20-25 weeks with weekly treatment sessions)/FUP (3 months post intervention)
  hair-cortisol concentrations (HCC) in the first 3 cm scalp hair segment at posterior vertex (~cumulative secretion over last 3 months)
Internalizing symptoms reported by the primary caregiver (CBCL) | pre-waitlist (before waiting period)/pre-treatment (within 3 weeks before start intervention)/mid-treatment (after 12 weeks with weekly treatment sessions)/post-treatment (after 20-25 weeks with weekly treatment sessions)/FUP (3 months post intervention)
  internalizing symptoms rated by primary caregivers using Child Behavior Checklist (CBCL 4-18). The scale ranges from 0-62 with higher scores indicating worse outcomes.
Internalizing symptoms reported by the secondary caregiver (CBCL) | pre-waitlist (before waiting period)/pre-treatment (within 3 weeks before start intervention)/mid-treatment (after 12 weeks with weekly treatment sessions)/post-treatment (after 20-25 weeks with weekly treatment sessions)/FUP (3 months post intervention)
  internalizing symptoms rated by primary caregivers using Child Behavior Checklist (CBCL 4-18). The scale ranges from 0-62 with higher scores indicating worse outcomes.
Quality of the parent-child interaction (EAS) | pre-waitlist (before waiting period) / pre-treatment (within 3 weeks before start of intervention), post-treatment (after 20-25 weeks with weekly treatment sessions) and follow up (3 months after intervention)
  In an exploratory fashion, the investigators will test whether the quality of parent-child interaction improve after the intervention and whether this improvement in interaction quality is a mediator of the treatment effect.
  Quality of the parent-child interaction assessed by the Emotional Availability Scales (EAS), specifically four caregiver scales (1. sensitivity, 2. structuring, 3. nonintrusiveness, and 4. nonhostility) and two child scales (1.responsiveness to mother and 2. involvement of mother). Codes on the scales range from 1 to 7, with higher scores indicating better outcome.
Quality of the parent-child interaction (MSSB) | pre-waitlist (before waiting period) / pre-treatment (within 3 weeks before start of intervention), post-treatment (after 20-25 weeks with weekly treatment sessions) and follow up (3 months after intervention)
  In an exploratory fashion, the investigators will test whether the child's ability to mentalize improve after the intervention and whether improvment in this ability is a mediator of the treatment effect.
  Child's ability to mentalize assessed by the Process Scales (Hill et al., 2009) MacArthur Narrative Coding Manual (MNCM; Robsinson et al., 2002) using the indices for narrative coherence (range: 1-12), intentionality (range: 1-12), with higher scores indicating better outcome.

OTHER OUTCOMES:
Feasibility-related endpoints - Acceptability of PaCT | post-treatment (after 20-25 weeks with weekly treatment sessions)
  Acceptability of PaCT rated by caregivers/ parents using Treatment evaluation questionnaire (FBB)
Feasibility-related endpoints - Acceptability of PaCT rated by children | post-treatment (after 20-25 weeks with weekly treatment sessions)
  Acceptability of PACT rated by children: Items derived from the German version of Therapeutic Alliance Scales for Children (TASC) assessed by Berkeley Puppet Interview technique (BPI)
Feasibility-related endpoints - Acceptability of PaCT rated by therapists | post-treatment (after 20-25 weeks with weekly treatment sessions)
  Acceptability of PaCT rated by therapists using Treatment evaluation questionnaire (FBB)
Feasibility-related endpoints - retention rates | post-treatment (after 20-25 weeks with weekly treatment sessions)
  Acceptability of PaCT: retention rates - the investigators expect a high rate of retention until post-treatment (expected 85%-90%)
Feasibility-related endpoints - adherence to PaCT | during all therapeutic sessions (20-25 weeks with weekly treatment sessions)
  Adherence to PACT interventions: coding of session videos using a Q-sort rating

CONTACTS AND LOCATIONS:
Overall Officials: Kai von Klitzing, Prof.Dr., Study Chair — University of Leipzig - Department of Child and Adolescent Psychiatry
Locations (1):
- University of Leipzig - Department of Child and Adolescent Psychiatry, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Yes
After publication of the primary objective, published data might be provided to interested scientists on request (e.g. for meta-analyses, health related registers or other scientific questions) in an anonymized way within 5 years, if the members of the TREAT-SAD-KIDS-trial group agree.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after publication within 5 years
Access Criteria: direct inquiry to coordinating investigators